CLINICAL TRIAL: NCT06057519
Title: Pragmatic Trial on the Safety and Tolerability of an Optimized Dose of Rifampicin in Tuberculosis Patients
Brief Title: Pragmatic Optimized Rifampicin Trial
Acronym: PORT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PORT- 01
Record Dates: First submitted 2023-08-07; First posted 2023-09-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized dose rifampicin (Experimental): 1800 mg flat dose
  Interventions: Drug: Optimised dose rifampicin
- Standard dose rifampicin (Active Comparator): 450 mg for patients under 50 kg and 600 mg for patients over 50 kg
  Interventions: Drug: Standard dose rifampicin

INTERVENTIONS:
Drug: Optimised dose rifampicin — Optimized dose of rifampicin
  Arms: Optimized dose rifampicin
Drug: Standard dose rifampicin — Standard dose rifampicin
  Arms: Standard dose rifampicin

SUMMARY:
The goal of this clinical trial is to compare an optimized dose (1800 mg) of rifampicin to standard dose (450 mg if patient <50 kg and 600 mg if patient >50kg) of rifampicin in tuberculosis patients.

The main questions it aims to answer are:

* To compare the incidence of hepatotoxicity occurs in the optimized dose vs standard dose arm
* To compare any adverse events occur in the optimized dose vs standard dose arm
* To compare final treatment outcome at the end of treatment according to WHO definitions of cure in the optimized dose regimen versus the standard dose regimen.
* To compare two and three months culture conversion rates in the optimized dose regimen versus the standard dose regimen.
* To describe and compare the steady-state plasma pharmacokinetics of the optimized dose regimen versus the standard dose regimen.

Participants will be given an optimized dose of 1800 mg of rifampicin daily. Researchers will compare the optimized and standard dose to see if more hepatotoxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* The patient has provided informed consent for study participation prior to all trial-related procedures.
* The patient has a diagnosis of pulmonary tuberculosis according to the local diagnostic criteria.
* The patient is aged 18 years or older at the day of informed consent.
* No known allergic reactions or toxicity to rifampicin in the past.
* Female patients of childbearing potential must have a negative serum pregnancy test, and consent to practice an effective method of birth control during the study. And they should not be lactating during the trial (female participants of childbearing potential only). Effective birth control for female patients has to include two methods, including methods that the patient's sexual partner(s) use. At least one must be a barrier method. Female patients are considered not to be of childbearing potential if they are post-menopausal with no menses for the last 12 months, or surgically sterile (this condition is fulfilled by bilateral oophorectomy, hysterectomy, and by tubal ligation which is done at least 12 months prior to enrolment).
* The patient will be compliant to the study schedule, in the discretion of the investigator.

Exclusion Criteria:

* The patient has tuberculosis which is assessed to receive high dose rifampicin according to the local standard of care.
* The patient started current TB treatment more than 4 weeks ago.
* The patient has TB meningitis.
* The patient is in a coma.
* Circumstances that raise doubt about free, uncoerced consent to study participation (e.g. in a prisoner or mentally handicapped person)
* The patient is not able to give consent personally.
* Poor general condition or comorbidities where delay in treatment cannot be tolerated or death within three months is likely. Or if there is concurrent treatment that may interfere.
* The patient is pregnant or breast-feeding.
* Patient infected with a rifampicin-resistant strain of M. tuberculosis.
* Known allergy or intolerance for rifamycins.
* The participant has a known or suspected, current alcohol or drug or amphetamine abuse, that is, in the opinion of the investigator, sufficient to compromise the safety or cooperation of the patient.
* The patient has a known allergy or intolerance, or concomitant disorders or conditions for which rifamycins or other standard TB treatment drugs are contraindicated.
* The patient has had treatment with any other investigational drug within 1 month prior to enrolment, or enrolment into other clinical (intervention) trials is planned in the upcoming 6 months
* Laboratory: at screening one or more of the following abnormalities were observed for the patient in screening laboratory:

  * Serum amino aspartate transferase (AST) and/or serum alanine aminotransferase (ALT) activity >3x the upper limit of normal
  * Serum total bilirubin level >2.5 times the upper limit of normal
  * Creatinine clearance (CrCl) level lower than 30 mls/min
* Acute or severe or life-threatening liver disease induced by drugs in the past
* The patient has a chronic disorder such as liver disease or renal disease.
* The patient has icterus.
* Previous anti-TB treatment: the patient ended a previous TB treatment (episode) within last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of hepatotoxicity | 26 weeks
  How often does hepatotoxicity occur in patients with optimized dose rifampicin vs standard dose rifampicin

SECONDARY OUTCOMES:
Adverse events | 26 weeks
  The proportion of adverse events overall and graded by severity assessed to be related or probably related to rifampicin will be compared between treatment arms.
Treatment outcome | 26 weeks
  Final treatment outcome at the end of treatment according to WHO definitions of cure will be compared between treatment arms
Culture conversion rate | 2 and 3 months post-treatment initiation
  Two and three months culture conversion rates will be compared between treatment arms.
PK parameter, AUC0-24 | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The AUC0-24 will be determined using sparse PK sampling.
PK parameter, Cmax | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The maximum concentration will be determined using sparse PK sampling.
PK parameter, Tmax | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The time to maximum concentration will be determined using sparse PK sampling.
PK parameter, Clearance | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The clearance of rifampicin will be determined using sparse PK sampling.
PK parameter, Volume of distribution | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The volume of distribution of rifampicin will be determined using sparse PK sampling.
PK parameter, T1/2 | 2 Weeks
  Steady-state plasma pharmacokinetic parameters will be compared between treatment arms. The half life of rifampicin will be determined using sparse PK sampling.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Boeree, Principal Investigator — Radboud University Medical Center
Locations (2):
- ASL Città di Torino, Turin, Italy
- Radboud University Medical Centre, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No